CLINICAL TRIAL: NCT04254029
Title: Short Term Cardiovascular and Renal Effects of Moringa Oleifera Extracts and Stevia Rebaudiana Bertoni as add-on Therapy in a Population of Type II Diabetes Individuals
Brief Title: The Cardiovascular and Renal Effects of Moringa Oleifera Extracts and Stevia Rebaudiana Bertoni in Patients With Type II Diabetes Mellitus
Acronym: MOROLSTEVER1
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Yaounde Central Hospital (Other Government)
Responsible Party: Principal Investigator, CN NGANOU-GNINDJIO, MD, MSc, Dr, Principal investigator, Yaounde Central Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MOROLSTEVER1
Record Dates: First submitted 2020-01-31; First posted 2020-02-05 (Actual); Last update posted 2020-02-05 (Actual); Status verified 2020-01

CONDITIONS: Benefits of a Capsules of Moringa Oleifera and Stevia Rebaudiana Bertoni in Patients With Type 2 Diabetes Mellitus Before and After 45 Days of add-on Therapy
Keywords: Diastolic function; Blood pressure profile; moringa oleifera; Stevia rebaudiana bertoni; Diabetes mellitus
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Non-randomized single-arm of MOROLSTEVER1 (Experimental): Non-randomized single-arm clinical trial with a before and after design. The study population consisted on all type 2 diabetes mellitus (T2DM) patients with a target population of T2DM patients with HbA1c between 42 to 64mmol/mol (6-8%) with no change in anti-diabetic treatment during the last three months, previous the study.
  The intervention consisted of a daily consummation of 425 ml of drink containing the extracts of 1,38mg of leaves extracts of moringa oleifera and 23,46 mg of stevia rebaudiana Bertoni leaves extracts lasting 45 days.
  Interventions: Dietary Supplement: MOROLSTEVER1

INTERVENTIONS:
Dietary Supplement: MOROLSTEVER1 — The intervention consisted of a daily consummation of 425 ml of drink containing the extracts of 1,38mg of leaves extracts of moringa oleifera and 23,46 mg of stevia rebaudiana Bertoni leaves extracts lasting 45 days.

SUMMARY:
The aim of the study was the evaluation of cardiovascular and renal benefits of moringa oleifera and stevia rebaudiana Bertoni in patients with type 2 diabetes mellitus before and after 8 weeks of add-on therapy.

DETAILED DESCRIPTION:
The investigators performed a non-randomized single-arm clinical trial with a before and after design, carried out from November 2016 and May 2017.

Intervention consisted of the administration of a daily consummation of 425 ml of drink containing the extracts of 1,38mg of leaves extracts of moringa oleifera and 23,46 mg of stevia rebaudiana Bertoni leaves extracts lasting 45 days. Before and after intervention, the following were done by the participants: bioelectrical impedance analysis (BIA), blood pressure measurements, fasting blood sugar, HbA1c, lipid profiles, liver function tests, kidney function tests, urinary excretion of albumin tests and full blood counts. These were followed by morphological workup including Electrocardiograms (ECGs), transthoracic heart ultrasounds and Ambulatory Blood Pressure Measurements (ABPM), also done before and after intervention.

Clinical evaluation with fasting blood sugar control, blood pressure controls and urinary excretion albumin tests were done for safety purposes.

ELIGIBILITY:
Inclusion Criteria:

* Known T2DM patients aged above 21years
* No change in anti-diabetic medication during the last three months HbA1c between 42 to 64mmol/mol (6-8%)
* Clearance of creatinine calculated according to the Modification of Diet in Renal Disease equation> 60ml/min/1.73 m2

Exclusion Criteria:

* Patient already on moringa or stevia supplementation or other herbal medication drugs that could interact with moringa or whose effects may be amplified, as far back as 1 month before study.
* Cardiac, renal disease and liver pathologies Sensitivity, intolerance or allergy to moringa or stevia Discontinued intervention
* Withdrawal of consent

Ages: 21 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Estimated)
Dates: Start 2016-11-01 (Actual); Primary Completion 2017-05-01 (Actual); Study Completion 2017-05-01 (Actual)

PRIMARY OUTCOMES:
Variation of mitral E' velocity | 45 days
  The mitral E' velocity is one of the methods for evaluating diastolic function.

SECONDARY OUTCOMES:
Variation of transmitral flow parameters such as E velocity | 45 days
  E (early diastolic filling velocity)
Urinary excretion of albumin | 45 days
  Urinary excretion of albumin level
Variation of blood pressure. | 45 days
  Change in systolic and diastolic blood pressure by using ABPM (mmHg)

CONTACTS AND LOCATIONS:
Locations (1):
- Yaounde Central Hospital, NAtional Obesity Center, Yaoundé, Cameroon